CLINICAL TRIAL: NCT04956692
Title: A Randomized, Phase 3, Open-label Study to Investigate the Pharmacokinetics and Safety of Subcutaneous Pembrolizumab Versus Intravenous Pembrolizumab, Administered With Platinum Doublet Chemotherapy, in the First-Line Treatment of Participants With Metastatic Squamous or Nonsquamous Non-Small-Cell Lung Cancer
Brief Title: Study of Pembrolizumab (MK-3475) Subcutaneous (SC) Versus Pembrolizumab Intravenous (IV) Administered With Platinum Doublet Chemotherapy in Participants With Metastatic Squamous or Nonsquamous Non-Small Cell Lung Cancer (NSCLC) (MK-3475-A86)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-A86; MK-3475-A86 (Other: MSD); jRCT2021210032 (Registry Identifier: jRCT (Japan Registry of Clinical Trials)); 2023-508308-40 (Registry Identifier: EU CT); U1111-1298-0215 (Other: UTN); 2020-002729-27 (EudraCT Number)
Record Dates: First submitted 2021-07-06; First posted 2021-07-09 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Programmed Cell Death 1 (PD1, PD-1); Programmed Cell Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death-Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Taxes; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy (Experimental): Participants receive pembrolizumab subcutaneous (SC) administration on Day 1 of each cycle (cycle length = 3 weeks) for up to 35 cycles (up to ~2 years) PLUS paclitaxel IV (on Day 1 of each cycle) OR nab-paclitaxel IV (on Days 1, 8, and 15 of each cycle) and carboplatin IV (on Day 1 of each cycle) for 4 cycles for squamous non-small cell lung cancer (NSCLC); PLUS carboplatin IV (on Day 1 of each cycle) Or cisplatin IV (on Day 1 of each cycle) for 4 cycles and pemetrexed IV (on Day 1 of each cycle) until progression, intolerable adverse events, or participant/physician decision for non-squamous NSCLC.
  Interventions: Biological: Pembrolizumab SC; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed
- Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy (Active Comparator): Participants receive pembrolizumab intravenous (IV) administration on Day 1 of each cycle (cycle length = 3 weeks) for up to 35 cycles (up to ~2 years) PLUS paclitaxel IV (on Day 1 of each cycle) OR nab-paclitaxel IV (on Days 1, 8, and 15 of each cycle) and carboplatin IV (on Day 1 of each cycle) for 4 cycles for squamous non-small cell lung cancer (NSCLC); PLUS carboplatin IV (on Day 1 of each cycle) Or cisplatin IV (on Day 1 of each cycle) for 4 cycles and pemetrexed IV (on Day 1 of each cycle) until progression, intolerable adverse events, or participant/physician decision for non-squamous NSCLC.
  Interventions: Biological: Pembrolizumab IV; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Biological: Pembrolizumab SC — SC injection
  Arms: Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy
Biological: Pembrolizumab IV — IV injection
  Other Names: MK-3475; KEYTRUDA®; SCH 900475
  Arms: Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Drug: Paclitaxel — IV injection
  Other Names: Nov-Onxol; Onxol; Paclitaxel Novaplus; Taxol
Drug: Nab-Paclitaxel — IV infusion
  Other Names: Abraxane; Nanoparticle albumin-bound paclitaxel
Drug: Carboplatin — IV infusion
  Other Names: Paraplatin; Paraplatin NovaPlus
Drug: Cisplatin — IV infusion
  Other Names: Platinol-AQ
Drug: Pemetrexed — IV infusion
  Other Names: LY231514; Alimta; Pemetrexed Disodium

SUMMARY:
The purpose of this study is to evaluate pembrolizumab (MK-3475) subcutaneous (SC) administration as the first-line therapy in the treatment of metastatic squamous and nonsquamous NSCLC by assessing the pharmacokinetics (PK), safety, and efficacy of pembrolizumab SC injection in combination with standard-of-care chemotherapy. The primary hypothesis of the study is Pembrolizumab SC is noninferior to pembrolizumab intravenous (IV) for Cycle 1 Area Under Curve (AUC) and Cycle 6 minimal concentration (Ctrough) at steady state.

Participants who discontinue study treatment after receiving the first course of 35 administrations of pembrolizumab (approximately up to 2 years) for reasons other than disease progression or intolerability, may be eligible for a second course of pembrolizumab for up to approximately 1 additional year if they have experienced radiographic disease progression per RECIST 1.1 as assessed by BICR after stopping first course treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has pathologically (histologically or cytologically) confirmed diagnosis of squamous or nonsquamous non-small cell lung cancer (NSCLC)
* Has Stage IV (T any, N any, M1a, M1b, or M1c - American Joint Committee on Cancer 8th Edition) squamous or nonsquamous NSCLC
* Has confirmation that epidermal growth factor receptor (EGFR), Anaplastic lymphoma kinase (ALK), or ROS Proto-Oncogene 1, Receptor Tyrosine Kinase (ROS1)-directed therapy is not indicated in nonsquamous NSCLC as well as mixed nonsquamous/squamous NSCLC. Participants with purely squamous NSCLC do not require testing
* Has not received prior systemic treatment for their metastatic NSCLC. Participants who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease
* Has an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0 or 1
* Male participants are eligible to participate if they agree to use contraception as per protocol unless confirmed to be azoospermic
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP) or is a WOCBP who agrees of using a contraceptive method per protocol
* Has measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by the local site investigator/radiology
* Submit an archival tumor tissue sample or newly obtained core or incisional biopsy of a tumor lesion not previously irradiated for PD-L1 status determination prior to randomization
* Has adequate organ function

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known central nervous system (ie, brain and/or spinal cord) metastases and/or carcinomatous meningitis. Participants with treated brain metastases may participate only if they satisfy all of the following: a) Have no evidence of new or enlarging brain metastases confirmed by post-treatment repeat brain imaging performed at least 4 weeks after pretreatment brain imaging, and b) Are neurologically stable without the need for steroids for at least 14 days before first dose of trial treatment as per local site assessment
* Has severe hypersensitivity to study intervention and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection and/or Hepatitis B infection or known active Hepatitis C infection
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has symptomatic ascites or pleural effusion. A participant who is clinically stable after treatment for these conditions is eligible
* Before the first dose of study intervention: a) Has received prior systemic cytotoxic chemotherapy for metastatic NSCLC b) Has received antineoplastic biological therapy for metastatic NSCLC c) Has had major surgery (<3 weeks prior to first dose) d) Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-programmed cell death ligand 2 (anti-PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Received radiation therapy to the lung that is >30 Gray within 6 months of the first dose of study intervention
* Is expected to require any other form of antineoplastic therapy while on study
* For participants with nonsquamous histology: Is unable to interrupt aspirin or other Non-steroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g/day, for a 5-day period
* For participants with nonsquamous histology: Is unable or unwilling to take folic acid or vitamin B12 supplementation
* Has received prior radiotherapy within 2 weeks of start of study intervention or have had a history of radiation pneumonitis. Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2026-10-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (126):
- United States (18):
  - St. Bernards Medical Center ( Site 0103), Jonesboro, Arkansas
  - St Joseph Heritage Healthcare-Oncology ( Site 0102), Fullerton, California
  - Cancer Blood and Specialty Clinic ( Site 0105), Los Alamitos, California
  - PIH Health Hematology Medical Oncology ( Site 0106), Whittier, California
  - Holy Cross Hospital ( Site 0017), Fort Lauderdale, Florida
  - Memorial Regional Hospital-Memorial Cancer Institute ( Site 0104), Hollywood, Florida
  - Advent Health ( Site 0013), Orlando, Florida
  - Fort Wayne Medical Oncology and Hematology ( Site 0101), Fort Wayne, Indiana
  - Baptist Health Lexington ( Site 0099), Lexington, Kentucky
  - St Luke's Hospital - Kansas City ( Site 0033), Kansas City, Missouri
  - St. Vincent Frontier Cancer Center ( Site 0058), Billings, Montana
  - Montefiore Medical Center [Bronx, NY] ( Site 0040), The Bronx, New York
  - The University of Tennessee Medical Center ( Site 0050), Knoxville, Tennessee
  - Tennessee Oncology ( Site 0051), Nashville, Tennessee
  - Oncology Consultants, PA ( Site 0052), Houston, Texas
  - Millennium Physicians - Oncology ( Site 0097), Houston, Texas
  - Oncology & Hematology Assoc. SW Virginia, Inc., DBA Blue Ridge Cancer Care ( Site 0100), Blacksburg, Virginia
  - West Virginia University ( Site 0056), Morgantown, West Virginia
- Brazil (5):
  - HOSPITAL EVANGÉLICO DE CACHOEIRO DE ITAPEMIRIM ( Site 0307), Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Sao Vicente de Paulo ( Site 0311), Passo Fundo, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia e Oncologia ( Site 0308), Joinville, Santa Catarina
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto ( Site 0305), São José do Rio Preto, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0304), São Paulo, São Paulo
- France (9):
  - Nouvel Hôpital Civil (NHC) ( Site 1018), Strasbourg, Bas-Rhin
  - CHU Limoges CHU Dupuytren ( Site 1011), Limoges, Haute-Vienne
  - Hôpital Foch ( Site 1019), Suresnes, Hauts-de-Seine
  - Institut Regional du Cancer de Montpellier - ICM ( Site 1003), Montpellier, Herault
  - Centre Hospitalier Sud Réunion ( Site 1020), Saint-Pierre, La Reunion
  - Hopital Guillaume & Rene Laennec ( Site 1007), Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier de Pau ( Site 1016), Pau, Pyrenees-Atlantiques
  - CHU de Rouen ( Site 1013), Rouen, Seine-Maritime
  - Hopital Cochin ( Site 1002), Paris
- Guatemala (5):
  - Centro de Investigaciones Clinicas de Latinoamerica S.A. - CELAN ( Site 0602), Guatemala City
  - Clinica Privada Dr. Rixci Ramirez ( Site 0601), Guatemala City
  - INTERVASC ( Site 0605), Guatemala City
  - Grupo Angeles SA ( Site 0604), Guatemala City
  - Centro Regional de Sub Especialidades Médicas SA ( Site 0600), Quetzaltenango
- Hungary (8):
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 1106), Kecskemét, Bács-Kiskun county
  - Petz Aladar Megyei Oktato Korhaz ( Site 1110), Győr, Győr-Moson-Sopron
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 1103), Szolnok, Jász-Nagykun-Szolnok
  - Tudogyogyintezet Torokbalint ( Site 1105), Törökbálint, Pest County
  - Veszprem Megyei Tudogyogyintezet ( Site 1108), Farkasgyepű, Veszprém megye
  - Zala Megyei Szent Rafael Korhaz ( Site 1111), Zalagerszeg, Zalaegerszeg
  - Semmelweis University-Pulmonológiai Klinika ( Site 1114), Budapest
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 1104), Budapest
- Japan (20):
  - Fujita Health University Hospital ( Site 3007), Toyoake, Aichi-ken
  - Ehime University Hospital ( Site 3005), Tōon, Ehime
  - Kurume University Hospital ( Site 3006), Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center ( Site 3014), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 3004), Kanazawa, Ishikawa-ken
  - Kanagawa Cardiovascular and Respiratory Center ( Site 3003), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 3000), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 3015), Sendai, Miyagi
  - Kurashiki Central Hospital ( Site 3013), Kurashiki, Okayama-ken
  - Kansai Medical University Hospital ( Site 3016), Hirakata, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 3009), Sakai, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 3017), Takatsuki, Osaka
  - Chiba University Hospital ( Site 3008), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 3001), Fukuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 3002), Fukuoka
  - Okayama University Hospital ( Site 3012), Okayama
  - Osaka International Cancer Institute ( Site 3018), Osaka
  - Tokushima University Hospital ( Site 3019), Tokushima
  - Juntendo University Hospital ( Site 3011), Tokyo
  - Showa University Hospital ( Site 3010), Tokyo
- Peru (6):
  - Hospital Nacional Carlos Alberto Seguin Escobedo ESSALUD ( Site 0704), Arequipa, Ariqipa
  - Clínica Peruano-Americana de Trujillo ( Site 0701), Trujillo, La Libertad
  - Oncosalud ( Site 0706), Lima, Muni Metro de Lima
  - Clinica Internacional Sede San Borja ( Site 0705), Lima
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 0703), Lima
  - Hospital Nacional Cayetano Heredia ( Site 0700), Lima
- Poland (6):
  - Przychodnia Lekarska KOMED ( Site 1202), Konin, Greater Poland Voivodeship
  - Centrum Onkologii im prof Franciszka Lukaszczyka ( Site 1201), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1206), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej ( Site 1205), Bystra, Silesian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 1200), Koszalin, West Pomeranian Voivodeship
- Romania (9):
  - Cardiomed SRL Cluj-Napoca ( Site 1313), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 1303), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL ( Site 1307), Comuna Floresti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 1304), Craiova, Dolj
  - Centrul de Oncologie Oncolab-Medical Oncology ( Site 1312), Craiova, Dolj
  - Spitalul Municipal Ploiesti ( Site 1308), Ploieşti, Prahova
  - Policlinica Oncomed SRL ( Site 1302), Timișoara, Timiș County
  - S.C.Focus Lab Plus S.R.L ( Site 1301), Bucharest
  - Spitalul Universitar de Urgenta Bucuresti ( Site 1305), Bucharest
- Russia (5):
  - SPBU Clinic of Advanced medical technologies n.a. N. I. Pirogov ( Site 1406), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 1407), Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg Scientific-Practical Center of Specialized Kinds of Medical Care (o) ( Site 1424), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary-Chemotherapy #1 ( Site 1425), Kazan', Tatarstan, Respublika
  - SPb SBHI City Clinical Oncological Dispensary ( Site 1409), Saint Petersburg
- South Africa (7):
  - Wits Clinical Research ( Site 1510), Johannesburg, Gauteng
  - Steve Biko Academic Hospital ( Site 1506), Pretoria, Gauteng
  - Marry Potter Oncology Centre ( Site 1502), Pretoria, Gauteng
  - Sandton Oncology Medical Group PTY LTD ( Site 1505), Sandton, Gauteng
  - Chris Hani Baragwanath Academic Hospital-Wits Clinical Research Bara ( Site 1513), Soweto, Gauteng
  - The Oncology Centre ( Site 1507), Durban, Limpopo
  - Cape Town Oncology Trials Pty Ltd ( Site 1500), Kraaifontein, Western Cape
- South Korea (3):
  - Chungnam National University Hospital ( Site 2002), Daejeon, Chungcheongnam-do
  - Chonnam National University Hwasun Hospital-Pulmonology ( Site 2000), Hwasun, Jeonranamdo
  - Korea University Guro Hospital ( Site 2003), Seoul
- Spain (5):
  - Hospital Insular de Gran Canaria-Oncology ( Site 1604), Las Palmas de Gran Canaria, Las Palmas
  - H.U. Vall de Hebron ( Site 1600), Barcelona
  - Hospital Juan Ramon Jimenez ( Site 1602), Huelva
  - Hospital Universitario Lucus Augusti ( Site 1603), Lugo
  - Hospital Universitario La Paz ( Site 1601), Madrid
- Taiwan (7):
  - Changhua Christian Hospital ( Site 2104), Changhua
  - National Taiwan University Hospital Hsin-Chu Branch ( Site 2103), Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 2107), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 2105), Tainan
  - National Taiwan University Hospital ( Site 2101), Taipei
  - Taipei Veterans General Hospital ( Site 2106), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 2102), Taoyuan District
- Turkey (Türkiye) (5):
  - Gulhane Egitim ve Arastirma Hastanesi ( Site 1704), Ankara
  - Ankara Sehir Hastanesi ( Site 1702), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1701), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 1703), Izmir
  - Inonu Universitesi Turgut Ozal Tip Merkezi ( Site 1707), Malatya
- Ukraine (8):
  - Medical Center Mriya Med-Service ( Site 1805), Kryvyi Rih, Dnipropetrovsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 1806), Kharkiv, Kharkivs’ka Oblast’
  - Ukrainian Center of Tomotherapy ( Site 1807), Kropyvnytskyi, Kirovohrad Oblast
  - Medical Center Asklepion LLC ( Site 1804), Khodosovka, Kyivska Oblast
  - Municipal non-profit enterprise'Odesa Regional Clinical Hosp-Thoracic surgery department. ( Site 181, Odesa, Odesa Oblast
  - Kremenchuk Regional Oncology Center ( Site 1811), Kremenchuk, Poltava Oblast
  - Kyiv City Clinical Oncology Centre ( Site 1809), Kyiv
  - Medical Center Dobrobut Clinic ( Site 1808), Kyiv

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26224&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Started | 358 | 173
Treated | 356 | 172
Completed | 0 | 0
Not Completed | 358 | 173
Not completed — Death | 115 | 47
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 2 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Ongoing in Study | 236 | 123

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy | Total
Number analyzed (Participants) | 358 | 173 | 531
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.6) | 65.6 (9.2) | 64.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 47 | 148
  Male | 257 | 126 | 383
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 27 | 77
  Not Hispanic or Latino | 307 | 146 | 453
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 72 | 32 | 104
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 232 | 113 | 345
  More than one race | 24 | 14 | 38
  Unknown or Not Reported | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cycle 1 Area Under The Curve From 0-3 Weeks (AUC 0-3wks) of Pembrolizumab
Description: Cycle 1 AUC0-3wks is defined as the area under the concentration-time curve for pembrolizumab in plasma over a 3-week dosing interval in Cycle 1. Each cycle is 21 days.
Time Frame: Cycle 1: predose and postdose day 1; days 2, 3, 4, 5, 6, 7, 10, and 15. Cycle 2: predose day 1. Each cycle is 21 days.
Population: The analysis population includes all randomized participants with at least 1 postdose sample in cycle 1, and for whom a model-based assessment could be done.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 355 | 170
hr*µg/mL | 471.33 [452.22 to 491.26] | 454.96 [438.54 to 471.99]
Statistical Analysis 1: Comparison: Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy vs Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy; Test type: Non-Inferiority — The non-inferiority margin with respect to the geometric means ratio (GMR) was 0.8; p < 0.0001, t-test, 1 sided — The one-sided p-value non-inferiority boundary is 0.02; Welch's unequal variances t-test. The null hypothesis was that GMR≤0.8; Geometric Mean Ratio (GMR) = 1.04, 96% CI 2-sided [0.98 to 1.10] — Numerator Arm A/Denominator Arm B

2. Primary Outcome: Cycle 6 Model-Based Minimal Concentration (Ctrough) of Pembrolizumab
Description: Cycle 6 model-based Ctrough is defined as the lowest concentration of pembrolizumab in plasma at the end of the dosing interval in Cycle 6, as predicted by the pharmacokinetic (PK) model based on historical intravenous pembrolizumab PK data. Each cycle is 21 days.
Time Frame: Cycle 6: predose day 1; days 2, 3, 4, 5, 6, 7, 10, and 15. Cycle 7: predose day 1. Each cycle is 21 days.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 240 | 93
µg/mL | 55.93 [53.05 to 58.96] | 30.25 [27.93 to 32.77]
Statistical Analysis 1: Comparison: Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy vs Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy; Test type: Non-Inferiority — The non-inferiority margin with respect to the geometric means ratio (GMR) was 0.8; p < 0.0001, t-test, 1 sided — The one-sided p-value non-inferiority boundary is 0.03; Welch's unequal variances t-test. The null hypothesis was that GMR≤0.8; Geometric Mean Ratio (GMR) = 1.85, 94% CI 2-sided [1.69 to 2.03] — Numerator Arm A/Denominator Arm B

3. Secondary Outcome: Objective Response (OR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: The OR rate is defined as the percentage of participants who achieve a confirmed complete response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2027-10

4. Secondary Outcome: Cycle 1 Observed Ctrough of Pembrolizumab
Description: Cycle 1 observed Ctrough is defined as the lowest observed concentration of pembrolizumab in plasma at the end of the dosing interval in Cycle 1. Each cycle is 21 days.
Time Frame: Predose Cycle 2 day 1. Each cycle is 21 days.
Population: The analysis population includes all randomized participants with at least 1 postdose sample in cycle 1.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 263 | 134
µg/mL | 18.36 [17.19 to 19.61] | 11.16 [10.49 to 11.88]

5. Secondary Outcome: Cycle 1 Maximum Concentration (Cmax) of Pembrolizumab
Description: Cycle 1 Cmax is defined as the observed peak concentration of pembrolizumab in plasma over the dosing interval in Cycle 1. Each cycle is 21 days.
Time Frame: Cycle 1: predose day 1; days 2, 3, 4, 5, 6, 7, 10, and 15. Cycle 2: predose day 1. Each cycle is 21 days.
Population: The analysis population includes all randomized participants with at least 1 postdose sample in cycle 1.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 355 | 170
µg/mL | 25.2 [23.8 to 26.6] | 58.3 [55.7 to 61.0]

6. Secondary Outcome: Cycle 6 AUC 0-3wks of Pembrolizumab
Description: Cycle 6 AUC0-3wks is defined as the area under the concentration-time curve for pembrolizumab in plasma over a 3-week dosing interval in Cycle 6. Each cycle is 21 days.
Time Frame: Cycle 6: predose and postdose day 1; days 2, 3, 4, 5, 6, 7, 10, and 15. Cycle 7: predose day 1. Each cycle is 21 days.
Population: The analysis population includes all randomized participants with at least 1 postdose sample in cycle 6, and for whom a model-based assessment could be done.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 240 | 93
hr*µg/mL | 1403.8 [1342.0 to 1468.5] | 952.9 [896.4 to 1013.0]

7. Secondary Outcome: Cycle 6 Cmax of Pembrolizumab
Description: Cmax in Cycle 6 is defined as the observed peak concentration of pembrolizumab in plasma over the dosing interval in Cycle 6. Each cycle is 21 days.
Time Frame: Cycle 6: predose and postdose day 1; days 2, 3, 4, 5, 6, 7, 10, and 15. Cycle 7: predose day 1. Each cycle is 21 days.
Population: The analysis population includes all randomized participants with at least 1 postdose sample in cycle 6.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 240 | 93
µg/mL | 65.6 [62.2 to 69.0] | 85.6 [80.1 to 91.4]

8. Secondary Outcome: Cycle 6 Observed Ctrough of Pembrolizumab
Description: Cycle 6 observed Ctrough is defined as the lowest observed concentration of pembrolizumab in plasma at the end of the dosing interval in Cycle 6. Each cycle is 21 days.
Time Frame: Predose Cycle 7 day 1. Each cycle is 21 days.
Population: The analysis population includes all randomized participants with at least 1 postdose sample in cycle 6.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 61 | 23
µg/mL | 57.17 [52.23 to 62.58] | 33.19 [29.53 to 37.30]

9. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be reported.
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted, anticipated posting 2027-10

10. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. The number of participants who discontinue study treatment due to an AE will be presented.
Time Frame: Up to approximately 25 months
Reporting Status: Not Posted, anticipated posting 2027-10

11. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by BICR
Description: PFS is defined as the time from randomization to the first documented PD per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2027-10

12. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2027-10

13. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR
Description: For participants who show confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, duration of response is defined as the time from the first documented evidence of CR or PR until disease progression (PD) per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2027-10

14. Secondary Outcome: Anti-Drug Antibodies (ADAs) Incidence After Administration of Pembrolizumab
Description: ADA incidence will be assessed by analyzing the development of ADAs following administration of pembrolizumab SC and pembrolizumab IV.
Time Frame: Up to approximately 26 months
Reporting Status: Not Posted, anticipated posting 2027-10

ADVERSE EVENTS:
Time Frame: Up to approximately 19 months
Description: All-Cause Mortality includes all participants who enrolled. Adverse Events include all participants who received ≥1 dose of study drug.
Arm/Group | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 118/358 | 48/173
Serious Adverse Events (participants affected / at risk) | 132/356 | 62/172
Other Adverse Events (participants affected / at risk) | 331/356 | 160/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy (N=356) | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy (N=172)
Anaemia (Blood and lymphatic system disorders) | 18 (19) | 2 (2)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (4)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Aplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 5 (5) | 3 (3)
Death (General disorders) | 3 (3) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Injection site exfoliation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 11 (11) | 10 (11)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyopneumothorax (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (2)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Pembrolizumab SC + Platinum Doublet Chemotherapy (N=356) | Arm B: Pembrolizumab IV + Platinum Doublet Chemotherapy (N=172)
Anaemia (Blood and lymphatic system disorders) | 188 (237) | 100 (118)
Neutropenia (Blood and lymphatic system disorders) | 116 (218) | 52 (107)
Thrombocytopenia (Blood and lymphatic system disorders) | 83 (137) | 40 (62)
Hyperthyroidism (Endocrine disorders) | 24 (26) | 7 (8)
Hypothyroidism (Endocrine disorders) | 25 (27) | 8 (8)
Constipation (Gastrointestinal disorders) | 57 (70) | 27 (33)
Diarrhoea (Gastrointestinal disorders) | 59 (77) | 23 (28)
Nausea (Gastrointestinal disorders) | 98 (141) | 48 (64)
Stomatitis (Gastrointestinal disorders) | 22 (24) | 5 (5)
Vomiting (Gastrointestinal disorders) | 32 (39) | 12 (17)
Asthenia (General disorders) | 46 (56) | 31 (38)
Fatigue (General disorders) | 41 (46) | 14 (15)
Oedema peripheral (General disorders) | 24 (25) | 13 (13)
Pyrexia (General disorders) | 24 (27) | 8 (8)
COVID-19 (Infections and infestations) | 24 (24) | 11 (11)
Alanine aminotransferase increased (Investigations) | 46 (60) | 26 (37)
Aspartate aminotransferase increased (Investigations) | 46 (63) | 29 (40)
Blood alkaline phosphatase increased (Investigations) | 18 (26) | 12 (14)
Blood creatinine increased (Investigations) | 34 (44) | 18 (27)
Blood lactate dehydrogenase increased (Investigations) | 22 (22) | 10 (11)
Lymphocyte count decreased (Investigations) | 19 (26) | 10 (15)
White blood cell count decreased (Investigations) | 50 (81) | 26 (41)
Decreased appetite (Metabolism and nutrition disorders) | 60 (74) | 25 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 24 (36) | 10 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 (20) | 12 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 17 (19) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (26) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (16) | 12 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (37) | 11 (19)
Dizziness (Nervous system disorders) | 17 (18) | 15 (17)
Headache (Nervous system disorders) | 20 (20) | 13 (15)
Neuropathy peripheral (Nervous system disorders) | 19 (21) | 8 (8)
Insomnia (Psychiatric disorders) | 22 (23) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 8 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 12 (13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 47 (47) | 23 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (27) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 25 (28) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT04956692/Prot_SAP_000.pdf